CLINICAL TRIAL: NCT02761148
Title: The Relationship Between White Matter Hyperintensity With Cognition and Emotion
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Minming Zhang, Chief,Department of Radiology,The 2nd Affiliated Hospital of Zhejiang University, School of Medicine, Zhejiang University
Other Study IDs: Z14H180003
Record Dates: First submitted 2016-05-02; First posted 2016-05-04 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Aged; Leukoaraiosis
Keywords: white matter hyperintensity; brain network; MRI; cognition; emotion
MeSH Terms: conditions — Leukoaraiosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Control
- White matter hyperintensity

SUMMARY:
White matter hyperintensity (WMH) has been found to be related with cognitive and emotional dysfunction. A presumed mechanism is that WMH disrupts the structural connectivity within a large-scale brain network, thereby impairing the brain's ability to integrate the neural processes efficiently. It is not yet clear, what the pattern of brain network disruption relates to WMH and how the brain network disruption induced by WMH has an effect on cognition and emotion performance. Using multi-model magnetic resonance imaging (MRI) techniques, we aimed to explore the mechanisms of cognitive decline and depression related with brain network dysfunction in patients with WMH, and to provide objective imaging marker for early diagnosis and prevention of WMH associated cognitive decline and depression.

ELIGIBILITY:
Inclusion criteria:

1. white matter hyperintensity visible on T2 fluid-attenuated inversion recovery images;
2. age between 35 to 80 years;
3. without stroke lesion (except lacunar infarction) on current diffusion weighted images;
4. without a history of multiple sclerosis, Alzheimer's disease, Parkinson's disease and head trauma.

Exclusion criteria:

1. white matter lesions of nonvascular origin (immunological-demyelinating, metabolic, toxic, infectious, other);
2. intracranial hemorrhage;
3. with severe head motion on magnetic resonance images

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: aged patients with white matter hyperintensity
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-01; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Fazekas Scale of white matter hyperintensity | 1 year
Mini-Mental State Examination (MMSE) | 1 year
Hamilton Depression Scale (HAMD) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- The 2nd Affiliated Hospital of Zhejiang University, School of Medicine,, Hangzhou, Zhejiang, China